CLINICAL TRIAL: NCT05364658
Title: A Clinical Evaluation of the Safety and Efficacy of the LensGen Intraocular Lens
Brief Title: A Clinical Evaluation of the LensGen Intraocular Lens
Acronym: Grail
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LensGen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LG-IOL-009
Record Dates: First submitted 2022-05-03; First posted 2022-05-06 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2022-05

CONDITIONS: Cataract; Presbyopia
MeSH Terms: conditions — Cataract; Presbyopia

STUDY DESIGN:
Intervention Model Description: Multi-center, open-label, non-comparative clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Juvene IOL (Experimental): Eyes that have been implanted with the LensGen Juvene IOL
  Interventions: Device: Juvene IOL

INTERVENTIONS:
Device: Juvene IOL — Indicated for Implantation in the human eye after removal of a cataractous crystalline lens

SUMMARY:
A multi-center, open-label, non-comparative clinical trial to assess the safety and efficacy of the LensGen IOL (Juvene IOL) for the treatment of aphakia and presbyopia after removal of the natural crystalline lens due to cataract.

DETAILED DESCRIPTION:
The Juvene IOL is specifically designed to utilize the mechanics of two optics to change the focal point in the human eye to correct presbyopia without the side effects experienced with other presbyopia correcting lenses. One optic provides the base power of the lens. The other contains a central fluid reservoir that utilizes the natural contraction of the ciliary body to change the focal point of the eye via the neural-uveal response induced by looking at an intermediate or near target.

The optic material is well characterized and has been safely used as an IOL material. Diffractive and refractive multifocal IOLs provide functional distance and near vision, with up to 4 diopters of add, yet they have not overcome the known side effects of haloes, glare, and reduced contrast sensitivity. Newer presbyopia correcting lenses, such as the Juvene IOL, use novel and proprietary changes in lens curvature to bilaterally change the focal point in each eye to any given distance the patient is looking.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 50 to 80 years
* In good general health at screening as determined by investigator
* Signed informed consent
* Cataract for which phacoemulsification extraction and posterior chamber IOL implantation has been planned
* Capsular bag size measured by UBM and determined to be a good fit for the Juvene IOL
* Preoperative best-corrected distance visual acuity (BCDVA) worse than 20/40 either with or without a glare source present (e.g., Brightness Acuity Tester), or scheduled for cataract removal due to significant cataract-related symptoms/complaints
* Calculated IOL power is within the range of the investigational IOL
* Preoperative "against the rule" corneal astigmatism (steep@180°) of 1.50 D or less or preoperative "with the rule" corneal astigmatism (steep @90°) of 0.75 D or less.
* Clear intraocular media other than cataract
* Availability, willingness, and sufficient cognitive awareness to comply with examination procedures
* Potential visual acuity of 20/32 or better in both eyes after cataract removal and IOL implantation as determined by diagnostic testing or investigator's judgement.
* No secondary procedures (such as LASIK) will be allowed during the term of the study

Exclusion Criteria:

* Uncontrolled systemic or ocular disease incuding clinically diagnosed significant dry eye syndrome (DES)
* Subjects taking medications that may affect ocular function (including but not limited t to mydriatic, cycloplegic and miotic agents; tricyclic antidepressants, phenothiazines, benzodiazepines, first generation antihistamines, and anticholinergic agents,)
* Systemic medications that may confound the outcome or increase the risk to the subject in the opinion of the investigator (tamsulosin hydrochloride (Flomax) or other medications with similar side effects (floppy iris syndrome))
* History of ocular trauma or prior ocular surgery
* Amblyopia or strabismus
* Any pathology that may affect visual acuity; particularly retinal changes that affect vision (macular degeneration, cystoid macular edema, proliferative diabetic retinopathy, glaucomatous optic neuropathy etc.)
* Keratoconus, pellucid corneal degeneration or other corneal dystrophy
* Irregular astigmatism
* Nystagmus
* Subjects who may be expected to require retinal laser treatment or other surgical intervention
* Capsule or zonular abnormalities that may affect postoperative lens stability (e.g.

pseudoexfoliation syndrome)

* Pupil abnormalities (non-reactive, tonic pupil, abnormally shaped pupil, rubeosis iridis, aniridia, or iris coloboma), or pupils that don't dilate at least 6.0 mm pharmacologically.
* Any pre-existing ocular conditions such as pseudoexfoliation, chronic uveitis, corneal dystrophy, traumatic cataract, white cataracts which lead to radicalization of the capsulorhexis
* Women who are pregnant or plan on getting pregnant during the term of the study
* Concurrent participation in another drug or device investigation
* Subjects shall be excluded when certain conditions are present at the time of surgery including:

  * Zonular instability
  * Need for iris manipulation
  * Capsular fibrosis or other opacity
  * Inability to fixate IOL in desired position

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2018-11-18 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Primary Effectiveness Endpoint | 12 Months
  Median, monocular, distance-corrected photopic intermediate visual acuity at 66cm is at least 0.2 logMar (20/32)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick R Casey, O.D., Study Director — LensGen, Inc.
Locations (2):
- Mexico (2):
  - Centro Oftamologico de Tijuana, Tijuana, Estado de Baja California
  - Dr. Enrique Barragan Oftalmologico, Monterrey, Nuevo León

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Garg S, De Jesus MT, Fletcher LM, Chayet A, Barragan E, Casey P. Twelve-month clinical outcomes after implantation of a new, modular, anterior shape-changing fluid optic intraocular lens. J Cataract Refract Surg. 2022 Oct 1;48(10):1134-1140. doi: 10.1097/j.jcrs.0000000000000935. PMID 35297798